CLINICAL TRIAL: NCT00374647
Title: Open Label Randomized Single Study to Evaluate the Safety & Efficacy of Early CNI Withdrawal in Recipients of Primary Renal Allografts Maintained Long-Term on Mycophenolate Mofetil; MMF (CellCept) and Sirolimus (Rapamune)
Brief Title: Study to Evaluate Safety and Efficacy of Early Calcineurin Inhibitor Withdrawal in Primary Renal Allografts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, E. Steve Woodle, Professor, University of Cincinnati
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STN INV INT
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Primary Renal Allograft
Keywords: Renal; Kidney; Transplant
MeSH Terms: interventions — Mycophenolic Acid; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: mycophenolate mofetil
Drug: sirolimus

SUMMARY:
Evaluate the safety and efficacy of early corticosteroid withdrawal and simultaneous calcineurin inhibitor withdrawal in recipients of primary renal allografts maintained long-term on MMF and sirolimus.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 75 years of age.
* Patients who are 90 to 240 days after having received a primary living or cadaver renal allograft.
* Patients maintained on a regimen of cyclosporine or tacrolimus and MMF since transplantation.
* Capable of providing written informed consent.
* No known contraindications to treatment with sirolimus.

Exclusion Criteria:

* Pregnant or lactating.
* Acute rejection within 90 days prior to study randomization.
* More than one biopsy proven acute rejection episode prior to study randomization.
* Previously received or are receiving an organ transplant other than kidney.
* Receiving sirolimus prior to entry.
* Severe diarrhea or other gastrointestinal disorders that may interfere with their ability to absorb oral medication.
* Evidence of active systemic infection requiring antibiotics, or HIV, HCV, HBV infection.
* History of malignancy in the past 5 years.
* Require dialysis at the time of study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of either acute rejection, biopsy proven calcineurin inhibitor toxicity, or failure of the estimated BSA indexed GFR by MDRD method to improve by 20% from time randomization to 12 months.

SECONDARY OUTCOMES:
Renal allograft function at 6 and 12 months.
Incidence of biopsy proven acute rejection at 6 and 12 months.
Time to first rejection.
Total number of rejection episodes per patient.
Graft loss and patient death.
Incidence of treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio